CLINICAL TRIAL: NCT00042965
Title: A Phase II Study Of Capecitabine Plus Gemcitabine For Metastatic Renal Cell Carcinoma
Brief Title: Capecitabine and Gemcitabine in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-90008; U10CA031946 (NIH); CDR0000069488 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2002-08-05; First posted 2003-01-27 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Kidney Cancer
Keywords: recurrent renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Capecitabine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine + capecitabine (Experimental): Patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15 and oral capecitabine twice daily on days 1-21. Treatment repeats every 28 days for a minimum of 2 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive at least 2 additional courses beyond CR.
  Patients are followed every 3 months for 1 year and then every 6 months for 1 year.
  Interventions: Drug: capecitabine; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: capecitabine
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining capecitabine with gemcitabine in treating patients who have metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response rate in patients with metastatic renal cell carcinoma treated with gemcitabine and capecitabine.
* Determine the duration of overall and progression-free survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed renal cell carcinoma

  * Clinically confirmed metastatic disease (histologic documentation of metastatic disease not required)
* Sarcomatoid renal cell carcinomas allowed
* No pure sarcomas
* No collecting duct (duct of Bellini) tumors, oncocytomas, or transitional cell tumors
* Measurable disease

  * At least 20 mm by conventional techniques OR
  * At least 10 mm by spiral CT scan
  * Nonmeasurable lesions include the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Lymphangitis cutis/pulmonis
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
* Patients with known brain metastases are eligible if they have undergone prior surgical resection and/or cranial irradiation, they currently do not require steroids or anticonvulsants, and there is no progressive disease on CT scan or MRI at least 4 weeks after completion of radiotherapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal

Renal

* Creatinine clearance at least 30 mL/min

Cardiac

* No clinically significant cardiac disease
* No congestive heart failure
* No symptomatic coronary artery disease
* No cardiac arrhythmias not well controlled with medication
* No myocardial infarction within the past 12 months

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 3 months after study
* No prior severe reaction to fluoropyrimidine therapy or known sensitivity to fluorouracil
* No malabsorption syndrome or lack of physical integrity of the upper gastrointestinal tract that would preclude absorption of capecitabine

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 4 weeks since prior chemotherapy and recovered
* No prior gemcitabine
* No prior fluoropyrimidines (e.g., fluorouracil, floxuridine, capecitabine, or fluorouracil-uracil)
* No other concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* At least 4 weeks since prior megestrol
* No concurrent hormones (e.g., megestrol) except steroids for adrenal failure, hormones for nondisease-related conditions (e.g., insulin for diabetes), or intermittent dexamethasone as an antiemetic

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered
* Prior radiotherapy to any lesion that may produce disability (e.g., unstable femur) allowed
* No concurrent palliative radiotherapy

Surgery

* See Disease Characteristics
* At least 4 weeks since prior major surgery and recovered

Other

* Any number of prior regimens allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2002-10; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Response rate | Up to 2 years

SECONDARY OUTCOMES:
Overall survival | Up to 2 years
Progression-free survival | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Walter M. Stadler, MD, FACP, Study Chair — University of Chicago
Locations (50):
- United States (49):
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Lifespan: The Miriam Hospital, Providence, Rhode Island
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Green Mountain Oncology Group, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
- McGill University, Montreal, Quebec, Canada

REFERENCES:
- [Result] Stadler WM, Halabi S, Rini B, Ernstoff MS, Davila E, Picus J, Barrier R, Small EJ; Cancer and Leukemia Group B. A phase II study of gemcitabine and capecitabine in metastatic renal cancer: a report of Cancer and Leukemia Group B protocol 90008. Cancer. 2006 Sep 15;107(6):1273-9. doi: 10.1002/cncr.22117. PMID 16909426
- [Result] Stadler WM, Halabi S, Ernstoff MS, et al.: A phase II study of gemcitabine (G) and capecitabine (C) in patients with metastatic renal cell cancer (mRCC): a report of Cancer and Leukemia Group B #90008. [Abstract] J Clin Oncol 22 (Suppl 14): A-4515, 385s, 2004.